CLINICAL TRIAL: NCT01402609
Title: A Randomized Controlled Trial Assessing the Efficacy of an Electronic Discharge Communication Tool for Preventing Death or Hospital Readmission
Brief Title: Assessing the Efficacy of an Electronic Discharge Communication Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ward of the 21st Century (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Health services (Other); University of Calgary (Other)
Responsible Party: Principal Investigator, William Ghali, Professor, Ward of the 21st Century
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SeamDis2010
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Other Diagnoses, Comorbidities, and Complications
Keywords: Continuity of care; Patient safety; Communication between acute and community care providers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group, usual care (Placebo Comparator): Control group will receive usual care. This usual care typically involves paper-based handwritten discharge communications, with subsequent provision of a dictated discharge summary produced some time after hospital discharge, with unpredictable success of delivery, and with unstructured and sometimes haphazard content.
  Interventions: Device: Usual care
- electronic discharge communication tool (Experimental): Patients allocated to the experimental arm will receive a copy of the discharge summary that is generated by the electronic discharge communication tool. The same copy is shared with their healthcare providers using an electronic, web-based, communication platform that allows communication between acute-care and community -care physicians. The electronic discharge communication tool allows physicians to start generating the discharge summary from time of admission to hospital.
  Interventions: Device: electronic discharge communication tool

INTERVENTIONS:
Device: electronic discharge communication tool — The intervention will consist of discharges being conducted with the use of the electronic discharge communication tool.For the intervention group, the care team will record the information that they collect directly into the computerized tool during the hospital stay.
  Other Names: seamless discharge
  Arms: electronic discharge communication tool
Device: Usual care — Control group will receive usual care. This usual care typically involves paper-based handwritten discharge communications, with subsequent provision of a dictated discharge summary produced some time after hospital discharge, with unpredictable success of delivery, and with unstructured and sometimes haphazard content.
  Other Names: dictation discharge
  Arms: Control group, usual care

SUMMARY:
The transition between acute care and community care represents one of the most vulnerable periods in health care delivery, particularly as the complexity of inpatient populations increases. Two recent North American studies found an incidence of post-discharge adverse events between 19-23%, with adverse drug events accounting for 66-72% of these. The vulnerability of this period has been attributed mainly to a failure of care providers to adequately reconcile discrepancies between home medications and discharge medications, as well as a failure to transfer this and other important information about the hospitalization and discharge to community care providers. While discharge communication with the primary care physician has traditionally occurred via a handwritten or dictated summary, major deficits exist with respect to timeliness of information transfer and adequacy of content in discharge summaries.

Computer-enabled discharge communications can potentially avert such problems. This is particularly true for web-based solutions that do not require end users to acquire additional software/training to use them. The purpose of this research is to definitively assess the efficacy of a web-based seamless discharge communication tool that the Medical Ward of the 21st Century (W21C - see www.w21c.org) team in Calgary has developed through iterative consultation with multiple clinical stakeholders as well as patients/families. This tool has great potential to be implemented on a provincial level as well as across Canada and internationally because it operates on a web interface that does not confine its applicability to a single type of hospital information system.

The purpose of this research is to definitively assess the efficacy of the web-based discharge communication tool that our team has developed in partnership with Alberta Health Services. In doing so, our specific objective will be to answer the following research questions:

1. Is the seamless discharge communication tool efficacious with respect to reducing hospital readmission and mortality (at 3 months), as well as reducing adverse events and adverse drug events?
2. Does the seamless discharge communication tool transfer appropriate, complete, and accurate discharge information in a timely manner compared to traditional discharge communication?
3. Is the seamless discharge communication tool efficacious with respect to improving physician and patient satisfaction?

DETAILED DESCRIPTION:
The vulnerability of the transition period has been attributed to three main factors. First, changes to patients'medication regimens during hospitalization are numerous, yet failure to reconcile discrepancies between admission and discharge is frequent. Second, the patient/family is required to take over care responsibilities at discharge and must often relay important information to the primary care physician. This can be particularly challenging if discharge information is poorly communicated, presented too rapidly, if instructions are verbal only, or if the patient has low literacy or low health literacy.Finally, crucial information is often not transferred between acute care physicians and community physicians.

Information about the hospitalization (such as medication changes, patient diagnoses, interventions,diagnostic findings, and necessary follow-up) is commonly transferred to the primary care physician via a discharge summary that is typically faxed or mailed. Unfortunately, deficits with respect to timeliness and/or complete failure to transmit are widespread. At the first post-discharge appointment, the discharge summary is unavailable to the primary care physician up to 75% of the time. This negatively impacts the continuity of care provided to many patients. When summaries are received, inconsistent content and inaccuracies are common. Acute care physicians, whether medical or surgical, often neglect to include diagnostic findings, treatment/hospital course, discharge medications, pending tests results, and whether the patient and family received counselling.

Computer-enabled discharge communications have potential to avert such problems. Such communication platforms can provide an immediate link between acute care and primary care physicians, and interfaces can be designed to ensure consistent information transfer. In addition, physicians in both settings have expressed preference for electronic discharge documents over hand written/dictated summaries with respect to clarity, comprehensiveness, and positive impacts on continuity of care.

ELIGIBILITY:
Inclusion Criteria:

* all patients being discharged from MTU at the Foothill Medical Centre (FMC)

Exclusion Criteria:

Patients will be excluded if the patient and/or family member decline consent; is under 18 years of age; cannot provide contact information; and/or family member lacks English proficiency and the team cannot communicate with them; has a research burden (enrolled in 2 other studies); is admitted under or has their acute care transferred to a clinical service other than the MTU; is not an Alberta resident; was previously enrolled in the study; is being discharged to hospice care; is transferred to another Hospital ("Rapid Transport"); is incoherent; or dies in hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1399 (Actual)
Dates: Start 2011-09; Primary Completion 2013-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
composite of death or readmission | 3 months
  The primary outcomes are identified as such because these are recognized to be major events that we are ultimately trying to prevent through safer health care. The 3 month time frame is felt to be most relevant, because it is short enough to potentially relate to discharge communications, but also long enough after discharge to permit some events to occur. The primary outcomes of interest will be assessed through existing linkages to hospitalization data from the Alberta Health Services Health Outcomes Group based in Calgary,for the outcome of readmission to acute care hospitals; and to data from Alberta Bureau of Vitals Statistics to determine all-cause mortality

SECONDARY OUTCOMES:
occurrence of post-discharge adverse events and adverse drug events at 1 month post discharge | 1 month post discharge

CONTACTS AND LOCATIONS:
Overall Officials: William Ghali, MD, Principal Investigator — Ward of the 21st Century
Locations (2):
- Canada (2):
  - Medical Teaching Unit, Foothills Medical Centre, Calgary, Alberta
  - The ward of 21st Century (W21C) Foothills Medical Centre, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kripalani S, Jackson AT, Schnipper JL, Coleman EA. Promoting effective transitions of care at hospital discharge: a review of key issues for hospitalists. J Hosp Med. 2007 Sep;2(5):314-23. doi: 10.1002/jhm.228. PMID 17935242
- [Background] van Walraven C, Seth R, Laupacis A. Dissemination of discharge summaries. Not reaching follow-up physicians. Can Fam Physician. 2002 Apr;48:737-42. PMID 12046369
- [Background] Callen JL, Alderton M, McIntosh J. Evaluation of electronic discharge summaries: a comparison of documentation in electronic and handwritten discharge summaries. Int J Med Inform. 2008 Sep;77(9):613-20. doi: 10.1016/j.ijmedinf.2007.12.002. Epub 2008 Feb 21. PMID 18294904
- [Background] van Walraven C, Laupacis A, Seth R, Wells G. Dictated versus database-generated discharge summaries: a randomized clinical trial. CMAJ. 1999 Feb 9;160(3):319-26. PMID 10065073
- [Derived] Sevick LK, Santana MJ, Ghali WA, Clement F. Prospective economic evaluation of an electronic discharge communication tool: analysis of a randomised controlled trial. BMJ Open. 2017 Dec 14;7(12):e019139. doi: 10.1136/bmjopen-2017-019139. PMID 29247110
- [Derived] Okoniewska BM, Santana MJ, Holroyd-Leduc J, Flemons W, O'Beirne M, White D, Clement F, Forster A, Ghali WA. The Seamless Transfer-of-Care Protocol: a randomized controlled trial assessing the efficacy of an electronic transfer-of-care communication tool. BMC Health Serv Res. 2012 Nov 21;12:414. doi: 10.1186/1472-6963-12-414. PMID 23170814
- See also: Research and Innovation centre located within the University of Calgary — http://www.w21c.org